CLINICAL TRIAL: NCT02215551
Title: Toward Optimizing Decompressive Laminectomy Outcomes: Looking Outside the Spine
Brief Title: Predictors of Decompressive Laminectomy Outcomes
Status: Completed | Type: Observational
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: O0798-R
Record Dates: First submitted 2014-07-22; First posted 2014-08-13 (Estimated); Last update posted 2023-01-12 (Actual); Status verified 2023-01

CONDITIONS: Lumbar Spinal Stenosis
Keywords: laminectomy
MeSH Terms: conditions — Spinal Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Study Group: Younger than 90 years old. no communication barriers (e.g., English speaking, household telephone) Affirmative response to each of the three following questions: a) Do patients have pain, weakness, numbness, or tingling in their legs when walking standing? b) Does this pain, weakness, numbness or tingling in their legs interfere with their daily activities? c) Have patients tried at least one non-surgical treatment for their leg symptoms (e.g., physical therapy, pain medications, spinal injection)? Have been scheduled for surgery on lower back for a condition called lumbar spinal stenosis.
  Whom have non degenerative causes of LSS such as tumor, infection, trauma, hemorrhage, or epidural lipomatosis, Prior lumbar spinal surgery, spondylolisthesis with spinal instability, significant cognitive impairment.

SUMMARY:
Decompressive laminectomy (DL) is the most common type of back surgery performed in older adults; DL treats lumbar spinal stenosis (LSS), a degenerative narrowing of the spinal canal causes pain and trouble walking. An estimated one in three people who undergo DL do not get well and often undergo repeated surgery.1,3-6 Some studies indicate that conditions outside of the spine (e.g., depression, hip arthritis) cause people who undergo DL to do poorly,27,30-36 but no one has comprehensively examined these conditions or the impact of treating them on DL outcomes. Thus LSS treatment continues to focus on the spine alone.61 The aim of this study is to identify conditions other than LSS that place Veterans at risk of poor DL outcomes so that future comparative effectiveness studies can be designed that examine the impact of a more comprehensive approach to treatment. Investigators believe that a patient-centered rather than a disease-centered approach will lead to superior outcomes, less suffering, and more appropriate use of health care resources.

DETAILED DESCRIPTION:
The primary aim of this 6-site prospective cohort study is to develop algorithms usable in the clinical setting that predict decompressive laminectomy (DL) outcomes (i.e., success vs. failure) in older adults with lumbar spinal stenosis (LSS), the most common indication for spine surgery in older patients. The clinical algorithms developed will be based primarily on factors outside of LSS that are important aging-related predictors of pain and disability (e.g., hip osteoarthritis (OA), fibromyalgia syndrome, depression, anxiety, fear-avoidance beliefs, dysfunctional coping). Preliminary data support the impact of some of these factors on DL outcomes, but no study has included comprehensive assessment of rigorously collected data in the context of a prospective cohort. Thus LSS treatment remains focused exclusively on the lumbar spine and treatment outcomes suboptimal with, on average, < 20% reduction in pain. An estimated one in three DL patients does not improve at all. Further, anatomical evidence of LSS (i.e., based on advanced imaging) exists in many older patients without pain or functional compromise. Two hundred fifty patients with symptomatic LSS scheduled to undergo DL without fusion and who have no dementia, spinal instability, or prior lumbar surgery will be recruited from spine surgery practices at each of the 6 participating sites (VA Pittsburgh Healthcare System, Durham VA Medical Center [MC], Richmond VAMC, Ann Arbor VAMC, Denver VAMC, San Antonio VAMC). Within 30 days prior to DL (i.e., at baseline), participants will undergo comprehensive and rigorous assessment of pain and disability-generating factors including: 1) SS symptoms with the Brigham Spinal Stenosis questionnaire (BSS, the most specific available LSS measurement tool); 2) musculoskeletal comorbidities (scoliosis, kyphosis, hip osteoarthritis, fibromyalgia symptoms, severity of spinal stenosis, degenerative disc and facet disease); 3) mood (depression [with the Centre for Epidemiology Studies Depression Scale (CES-D)], anxiety [with the GAD-7]); 4) cognitive function (normal vs. mild cognitive impairment with the computer-based assessment of mild cognitive impairment); 5) psychological function (fear-avoidance beliefs [with the Fear Avoidance Beliefs Questionnaire], chronic pain self-efficacy [with the Chronic Pain Self-Efficacy Scales], dysfunctional pain coping skills [with the Cognitive Strategies Questionnaire], treatment expectancy, illicit substance use, alcohol use, smoking status, PTSD symptoms); 6) medical comorbidity (including BMI); 7) demographic factors (age, gender, race, educational/marital status). The BSS will be collected at baseline, at the first postoperative visit, and every 3 months for one year. Prediction rules, based on the comprehensive set of factors measured and DL success/failure determined by the BSS, will be created using multiple methods to maximize predictive accuracy and validated subsequently in a separate cohort of 100 individuals. Investigators will apply these rules to future comparative effectiveness trials that test personalized LSS treatment approaches (i.e., that involve targeting extra-LSS factors as part of the total treatment package) as compared with DL alone. An exploratory aim of the proposed study is to evaluate the use of Goal Attainment Scaling (GAS) as a DL outcome. This patient-centered outcomes measurement approach is used commonly in the rehabilitation setting, but never before in DL patients. To prepare for future comparative effectiveness trials, investigators want to develop GAS as an outcome measure because it can be used to track outcomes in SS patients across surgical and non-surgical interventions, and investigators anticipate that both will be employed as part of personalized treatment. Investigators will explore (through 10-12 patient interviews) and refine (with a modified Delphi panel of experts) GAS goals in patients with SS, and measure goal achievement in a subset of 20 participants. What might happen if older adults with LSS were treated in the context of a comprehensive pre-operative program before undergoing DL? Might long-term outcomes associated with DL improve? Might patient satisfaction improve? Might some patients avoid DL? These are questions that ultimately investigators hope to answer.

ELIGIBILITY:
Inclusion Criteria:

* Younger than 90 years old.
* no communication barriers (e.g., English speaking, household telephone)
* Affirmative response to each of the three following questions:

  * a) Do patients have pain, weakness, numbness, or tingling in their legs when walking standing?
  * b) Does this pain, weakness, numbness or tingling in their legs interfere with their daily activities?
  * c) Have patients tried at least one non-surgical treatment for their leg symptoms (e.g., physical therapy, pain medications, spinal injection)?
* Have been scheduled for surgery on lower back for a condition called lumbar spinal stenosis.

Exclusion Criteria:

* non degenerative causes of LSS such as

  * tumor,
  * infection,
  * trauma,
  * hemorrhage,
  * or epidural lipomatosis
* Prior lumbar spinal surgery
* spondylolisthesis with spinal instability
* significant cognitive impairment

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 350 Veterans with degenerative lumbar spinal stenosis (LSS) who are scheduled to undergo decompressive laminectomy (DL) will be recruited. No one will be excluded on the basis of age, race, gender or ethnicity. There is no age restriction as investigators are targeting patients with degenerative lumbar spinal stenosis, most of who are in their 50's and 60's. Investigators exclude participants with non-degenerative causes of LSS, as noted below. Investigators anticipate that the demographics of the participants will reflect that of the three participating VA sites and their affiliated University spine surgery practices. Our goal is to recruit at least 70% Veteran participants and Investigators have added three additional VA sites that will help to ensure this.
Sampling Method: Non-Probability Sample
Enrollment: 239 (Actual)
Dates: Start 2014-10-01 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2023-01-10 (Actual)

PRIMARY OUTCOMES:
Brigham Spinal Stenosis Questionnaire | 1 Year
  The BSS has three scales that measure pain, function, and satisfaction. The pain and satisfaction scales can be administered before and after DL; the satisfaction scale measures satisfaction with surgery and is only administered following DL. Threshold values have been defined for success versus failure on each of the three subscales based on receiver operating characteristic (ROC) analyses - 0.46 for the Symptom Severity Scale, 0.42 for the Physical Function Scale, and 2.42 for the Patient Satisfaction Scale. The most balanced definition of overall success requires that the patient achieve success in at least two of the three scales. Investigators use this definition, which has the greatest sensitivity and specificity, as the primary outcome in our statistical analyses.

OTHER OUTCOMES:
Goal Attainment Scaling (GAS) | 1 Year
  Goal Attainment Scaling is a structured interview that allows for standardized measurement of physical function goals in terms of the degree to which they have been attained for each individual person.

CONTACTS AND LOCATIONS:
Overall Officials: Debra K. Weiner, MD, Principal Investigator — VA Pittsburgh Healthcare System University Drive Division, Pittsburgh, PA
Locations (7):
- United States (7):
  - VA Eastern Colorado Health Care System, Denver, CO, Denver, Colorado
  - Atlanta VA Medical and Rehab Center, Decatur, GA, Decatur, Georgia
  - VA Ann Arbor Healthcare System, Ann Arbor, MI, Ann Arbor, Michigan
  - Minneapolis VA Health Care System, Minneapolis, MN, Minneapolis, Minnesota
  - VA Pittsburgh Healthcare System University Drive Division, Pittsburgh, PA, Pittsburgh, Pennsylvania
  - South Texas Health Care System, San Antonio, TX, San Antonio, Texas
  - Hunter Holmes McGuire VA Medical Center, Richmond, VA, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No